CLINICAL TRIAL: NCT05930080
Title: Multi-center, Randomized, Double Blinded, Active-controlled Phase III Clinical Trial to Assess the Efficacy and Safety of SKCPT in Patients With Knee Osteoarthritis
Brief Title: Efficacy and Safety of SKCPT in Patients With Knee Osteoarthritis: Phase III Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKCPT_001
Record Dates: First submitted 2023-06-20; First posted 2023-07-05 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKCPT group (Experimental)
  Interventions: Drug: SKCPT
- Celebrex group (Active Comparator)
  Interventions: Drug: Celebrex

INTERVENTIONS:
Drug: SKCPT — the randomly assigned subjects took the study drug for 12 weeks
  Arms: SKCPT group
Drug: Celebrex — the randomly assigned subjects took the study drug for 12 weeks
  Arms: Celebrex group

SUMMARY:
Multi-center, Randomized, Double Blinded, Active-controlled Phase III Clinical Trial to Assess the Efficacy and Safety of SKCPT in Patients with knee Osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 20 to 75 years
* Kellgren-Lawrence (KL) grade 1 to 3
* Individuals who voluntarily decide to participate in the study and provide written informed consent form
* Individuals who can understand and follow instructions and can participate in the study during the entire study period

Exclusion Criteria:

* Individuals who have clear secondary osteoarthritis caused by inflammatory, infectious, metabolic arthritis, or other conditions such as rheumatoid arthritis, rather than primary knee osteoarthritis as determined by the investigator
* Individuals with other factors that could potentially affect the assessment of this clinical study due to pain caused by osteoarthritis or other conditions in the hip joint
* Individuals who have undergone knee joint arthroplasty
* Individuals who have undergone open knee surgery (ligament reconstruction, osteotomy) within 3 years prior to the screening visit

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
K-WOMAC Pain Subscale | 84 days
  The average changes in the K-WOMAC(Western Ontario and McMasters Universitis) Pain Subscale (range: 0-100 mm, higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No